CLINICAL TRIAL: NCT04368767
Title: A Pilot Randomized Controlled Trial of the Effects of Daily Skin-to-skin Contact Compared to Standard Care on the Stress Responses of Late Preterm Infants in the First Week of Life
Brief Title: A Pilot Randomized Controlled Trial of the Effects of Daily Skin-to-skin Contact (PRCTS2S)
Acronym: PRCTS2S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-29543
Record Dates: First submitted 2019-11-26; First posted 2020-04-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Premature Baby 33 to 36 Weeks; Mother-Infant Interaction; Oxidative Stress

STUDY DESIGN:
Intervention Model Description: We will use a randomized controlled trial design to examine feasibility of the prolonged SSC intervention in the first week of life for late preterm infants and to provide preliminary data for future research to compare the effects of usual incubator care with prolonged SSC on biomarkers of stress in late preterm infants in the first week of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care: Incubator (No Intervention): The infant will remain in the incubator and stress biomarkers will be collected per protocol
- Intervention: Skin-to-skin (Experimental): Skin-to-skin contact will be performed for two hours daily for three consecutive days in the first week of life, 30 minutes after feeding. SSC will usually occur in the afternoon between 11:30-12:30 pm or 14:30-15:30pm. This time interval will allow all pre-intervention sample collection to begin 1 hour after the infant's feeding schedule in the afternoon. The room will be monitored to maintain a temperature of 72-77 degrees Fahrenheit during SSC. Stress biomarkers will be collected per protocol.
  Interventions: Behavioral: Skin-to-skin

INTERVENTIONS:
Behavioral: Skin-to-skin — Skin-to-skin contact will be performed for two hours daily for three consecutive days in the first week of life, usually in the afternoon. This time interval will allow all pre-intervention sample collection to begin 1 hour after the infant's feeding schedule in the afternoon. After pre-intervention measures of axillary temperature, heart rate, respiratory rate, and oxygen saturation by pulse oximetry (SPO2) are obtained; cotton balls placed in the diaper for urine collection will be removed and stored in an appropriate container. Salivary oxytocin and cortisol will be collected per protocol below. Mothers will be requested to sit in reclining chairs with a front opened blouse or hospital gown. Infants will be removed from the incubator and placed naked except for a diaper and hat directly onto the skin between the mother's breasts and covered with a blanket. All infants will be monitored. After the two hours of SSC is completed, the infant will be returned to the incubator.
  Arms: Intervention: Skin-to-skin

SUMMARY:
Late preterm infants are at risk of experiencing inadequate glycogen stores with immature glucose metabolism and increased adenosine triphosphate (ATP) degradation, which indicates cellular increased and stress. Processes mediating infant acute/chronic stress symptoms and their biochemical effects have not been adequately investigated. Skin-to-skin contact (SSC), also known as Kangaroo Mother Care (KMC), is as an intervention that activates mechanisms of energy preservation that decrease stress in preterm infants. SSC has been shown in numerous clinical trials to reduce mortality and morbidity by stabilization of breathing, thermal regulation, oxygen saturation, and heart rate. SSC also reduces behavioral distress during painful and stressful procedures and improves breast-feeding parent bonding. However, little is known about how SSC affects biomarkers of stress and energy expenditure in late preterm infants in the first week of life.

The aim of this pilot randomized controlled trial is to evaluate changes in biomarkers of stress, stress modulation and energy expenditure in late preterm infants who receive two hours of continuous SSC care or two hours of lying undisturbed in an incubator administered daily for 3 consecutive days in the first week of life, and to provide preliminary data for future research comparing the effects of usual incubator care with prolonged SSC on stress biomarkers in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 34 weeks and 0/7 days through 35 weeks and 6/7 days gestational age
* Medically stable as determined by a Neonatal Acute Physiology- Perinatal Extension SNAPPE -II (SNAPPE-II) score of less than 9
* Mothers able to read and write English
* Mothers have no medical contraindications to holding their infant in SSC for up to 2 hours

Exclusion Criteria:

* Surgery in the first week of life
* Intraventricular hemorrhage (IVH) of grade 3 or 4
* Opioids, benzodiazepines, muscle relaxants, phenobarbital, and/or dilantin
* Plasma creatinine of >1 mg/dl
* Severe cyanotic heart disease or severe respiratory distress
* Abdominal wall or intestinal anomaly or injury (NEC)
* Facial anomaly or other known chromosomal anomaly
* Life-threatening congenital anomaly or are so critically ill that they are unlikely to survive or are receiving palliative care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Preterm Infants - not gender based Mothers of preterm infants - gender based
Enrollment: 8 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Stress biomarkers | Day 3
  Compare group differences in measures of stress (i.e., salivary cortisol, urinary biomarkers of Hx, Xa, UA, and allantoin, and stress buffering (i.e., salivary oxytocin) between the intervention and usual care groups.
Stress biomarkers | Day 2
  Compare group differences in measures of stress (i.e., salivary cortisol, urinary biomarkers of Hx, Xa, UA, and allantoin, and stress buffering (i.e., salivary oxytocin) between the intervention and usual care groups.
Stress biomarkers | Day 1
  Compare group differences in measures of stress (i.e., salivary cortisol, urinary biomarkers of Hx, Xa, UA, and allantoin, and stress buffering (i.e., salivary oxytocin) between the intervention and usual care groups.

SECONDARY OUTCOMES:
Mother's Satisfaction with SSC | Day 3
  Mother's Satisfaction with SSC Questionnaire
Number of discomforting and stressful events for mother | Day 3
  Total count of discomfort and stressful events
Number of discomforting and stressful events for mother | Day 2
  Total count of discomfort and stressful events
Number of discomforting and stressful events for mother | Day 1
  Total count of discomfort and stressful events
Number of discomforting and stressful events for infant | Day 3
  Total count of discomforting and stressful events
Number of discomforting and stressful events for infant | Day 2
  Total count of discomforting and stressful events
Number of discomforting and stressful events for infant | Day 1
  Total count of discomforting and stressful events
Change in stress biomarkers | pre and post the intervention on days 1, 2, and 3
  salivary cortisol, urinary biomarkers of Hx, Xa, Uric Acid (UA), and allantoin and stress buffering (i.e., salivary oxytocin

CONTACTS AND LOCATIONS:
Overall Officials: Linda Franck, RN, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Isayama T, Lewis-Mikhael AM, O'Reilly D, Beyene J, McDonald SD. Health Services Use by Late Preterm and Term Infants From Infancy to Adulthood: A Meta-analysis. Pediatrics. 2017 Jul;140(1):e20170266. doi: 10.1542/peds.2017-0266. PMID 28759410
- [Result] Blass E. Energy conservation in infants. Behav Processes. 2015 Aug;117:35-41. doi: 10.1016/j.beproc.2015.01.011. Epub 2015 Jan 30. PMID 25643950
- [Result] Tan JBC, Boskovic DS, Angeles DM. The Energy Costs of Prematurity and the Neonatal Intensive Care Unit (NICU) Experience. Antioxidants (Basel). 2018 Mar 2;7(3):37. doi: 10.3390/antiox7030037. PMID 29498645
- [Result] Chi Luong K, Long Nguyen T, Huynh Thi DH, Carrara HP, Bergman NJ. Newly born low birthweight infants stabilise better in skin-to-skin contact than when separated from their mothers: a randomised controlled trial. Acta Paediatr. 2016 Apr;105(4):381-90. doi: 10.1111/apa.13164. Epub 2015 Oct 15. PMID 26303808
- [Result] Morelius E, He HG, Shorey S. Salivary Cortisol Reactivity in Preterm Infants in Neonatal Intensive Care: An Integrative Review. Int J Environ Res Public Health. 2016 Mar 18;13(3):337. doi: 10.3390/ijerph13030337. PMID 26999185
- [Result] Kim KM, Henderson GN, Ouyang X, Frye RF, Sautin YY, Feig DI, Johnson RJ. A sensitive and specific liquid chromatography-tandem mass spectrometry method for the determination of intracellular and extracellular uric acid. J Chromatogr B Analyt Technol Biomed Life Sci. 2009 Jul 15;877(22):2032-8. doi: 10.1016/j.jchromb.2009.05.037. Epub 2009 May 27. PMID 19520625
- [Result] Tolun AA, Zhang H, Il'yasova D, Sztaray J, Young SP, Millington DS. Allantoin in human urine quantified by ultra-performance liquid chromatography-tandem mass spectrometry. Anal Biochem. 2010 Jul 15;402(2):191-3. doi: 10.1016/j.ab.2010.03.033. Epub 2010 Mar 31. PMID 20361921
- [Result] Cong X, Ludington-Hoe SM, Hussain N, Cusson RM, Walsh S, Vazquez V, Briere CE, Vittner D. Parental oxytocin responses during skin-to-skin contact in pre-term infants. Early Hum Dev. 2015 Jul;91(7):401-6. doi: 10.1016/j.earlhumdev.2015.04.012. Epub 2015 May 16. PMID 25988992
- [Result] Plank MS, Calderon TC, Asmerom Y, Boskovic DS, Angeles DM. Biochemical measurement of neonatal hypoxia. J Vis Exp. 2011 Aug 24;(54):2948. doi: 10.3791/2948. PMID 21897351